CLINICAL TRIAL: NCT07340112
Title: Expression of GLP1 Receptor on Peripheral Blood Mononuclear Cells in Advanced Peripheral Artery Disease: Paving the Way for GLP1R Agonists Treatment in Chronic Limb Threatening Ischemia
Acronym: EXCEL-CLTI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Centre de Recherche en biomédecine de Strasbourg INSERM UMR-S1118 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 9908
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease (PAD); Claudication, Intermittent; Chronic Limb-Threatening Ischemia
Keywords: Peripheral arterial disease; Chronic limb-threatening ischemia; GLP-1 receptor; Peripheral blood mononuclear cells (PBMC)
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample (15 mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Limb-Threatening Ischemia (CLTI): A group of patients presenting with chronic limb-threatening ischemia, the most severe form of peripheral artery disease
  Interventions: Diagnostic Test: Analysis of GLP-1 receptor expression
- Intermittent claudication (IC): A group of patients presenting with intermittent claudication, a less advanced stage of of peripheral artery disease, serving as a comparator
  Interventions: Diagnostic Test: Analysis of GLP-1 receptor expression

INTERVENTIONS:
Diagnostic Test: Analysis of GLP-1 receptor expression — One-time 15mL blood sampling for GLP-1R expression analysis on PBMCs via RT-qPCR and Western blot

SUMMARY:
The goal of this observational study is to learn whether activation of the GLP-1 receptor could represent a therapeutic target by characterizing its expression and associated inflammatory mechanisms in patients with peripheral artery disease, according to disease severity, in adults with symptomatic lower-limb peripheral arterial disease.

The main questions it aims to answer are:

* Is the level of GLP-1 receptor (GLP1R) expression on peripheral blood mononuclear cells (PBMC) different between patients with intermittent claudication (ischemia of effort) and those with chronic limb-threatening ischemia?
* Is GLP1R expression associated with inflammatory and oxidative profiles of PBMC?
* Can GLP-1 receptor agonists reverse inflammatory and oxidative alterations induced by plasma from patients with peripheral artery disease in endothelial cell cultures?
* Are there specific plasma proteomic signatures associated with GLP1R overexpression?

Researchers will compare patients with intermittent claudication to patients with chronic limb-threatening ischemia to see if disease severity is associated with differences in GLP1R expression, PBMC inflammatory/oxidative phenotype, and plasma proteomic profiles.

Participants will:

* Provide an additional blood sample (15 mL) collected during a routine, clinically indicated blood draw
* Have PBMC isolated for measurement of GLP1R expression and assessment of inflammatory and oxidative markers
* Have plasma analyzed for proteomic profiling and used in in-vitro endothelial cell experiments

Participation ends after completion of the blood sampling, and no additional procedures beyond standard clinical care are required.

DETAILED DESCRIPTION:
Chronic limb-threatening ischemia is the most severe stage of lower-limb peripheral arterial disease and remains associated with poor cardiovascular and limb prognosis. This condition is characterized by a pronounced systemic inflammatory and oxidative state, in which peripheral blood mononuclear cells play a central role.

Glucagon-like peptide-1 receptor agonists have shown anti-inflammatory and cardiovascular protective effects in other settings, but the involvement of the GLP-1 receptor in severe peripheral arterial disease has not been clearly established. This pilot study aims to characterize GLP-1 receptor expression on peripheral blood mononuclear cells according to disease severity and to evaluate its association with inflammatory, oxidative, and proteomic profiles.

This is a monocentric, cross-sectional observational study conducted at the CHU of Strasbourg. Patients hospitalized for evaluation of symptomatic lower-limb peripheral arterial disease will be classified into intermittent claudication or chronic limb-threatening ischemia groups. A single additional blood sample will be collected during routine clinical sampling. Peripheral blood mononuclear cells and plasma will be analyzed to assess GLP-1 receptor expression, inflammatory and oxidative markers, and plasma proteomic signatures. Exploratory in-vitro experiments will evaluate the ability of GLP-1 receptor agonists to reverse endothelial alterations induced by patient plasma.

The study is designed to generate mechanistic data supporting the GLP-1 receptor as a potential therapeutic target in chronic limb-threatening ischemia and to inform future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older
* Documented Peripheral Artery Disease (PAD): Patients must fall into one of the two following severity groups:

  1. Intermittent Claudication (IC) Group: Defined by a maximum walking distance limited by intermittent claudication, associated with an Ankle-Brachial Index (ABI) < 0.9 at rest.
  2. Chronic Limb-Threatening Ischemia (CLTI) Group: Defined by ischemic rest pain and/or tissue loss (ulcers or gangrene) persisting for at least 15 days, associated with a toe pressure or a transcutaneous oxygen tension (tcPO2) < 30 mmHg, according to the 2024 ESC guidelines.

Exclusion Criteria:

* Diabetes Mellitus: Diagnosis of Type 1 or Type 2 diabetes
* Current Specific Pharmacotherapy: Ongoing treatment with SGLT2 inhibitors (SGLT2i) or GLP-1 receptor agonists (GLP-1RA).
* Infection: Presence of sepsis or an active systemic infection.
* Malignancy: Active cancer or hematologic malignancies.
* Immunosuppression: History of organ transplantation or autoimmune diseases currently requiring immunosuppressive therapy.
* Known chronic inflammatory diseases.
* Advanced Renal Failure: End-stage renal disease requiring dialysis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the patient population managed at the Strasbourg University Hospital (CHU de Strasbourg), France. The cohort consists of individuals referred to the vascular surgery and vascular medicine departments for specialized tertiary care. Participants are identified and enrolled during their scheduled medical or surgical hospitalizations, including both outpatient day-hospital units and conventional inpatient wards. The population represents a real-world clinical sample of symptomatic patients undergoing standardized diagnostic or therapeutic evaluations for peripheral arterial conditions.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Level of GLP-1 Receptor (GLP-1R) Gene Expression in PBMCs | Day 1 (at the time of the one-time blood sampling)
  Quantification of GLP-1R mRNA expression levels in Peripheral Blood Mononuclear Cells (PBMCs) using RT-qPCR. This measure aims to compare the level of receptor expression between patients with Intermittent Claudication and those with Chronic Limb-Threatening Ischemia.

SECONDARY OUTCOMES:
Systemic Pro-inflammatory Cytokine Profile | Day 1
  Concentration of pro-inflammatory cytokines (IL-1β, IL-6, and TNF-α) measured in pg/mL using ELISA
Oxidative and Nitrosative Stress Markers in PBMCs | Day 1
  Measurement of Nitric Oxide (NO) and Reactive Oxygen Species (ROS) levels in PBMCs using fluorescent probes and flow cytometry (expressed as Mean Fluorescence Intensity).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No